CLINICAL TRIAL: NCT02224768
Title: YERVOY Risk Minimisation Tool Evaluation Survey
Brief Title: YERVOY® Risk Minimization Tool Effectiveness Evaluation Survey
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-242
Record Dates: First submitted 2014-03-20; First posted 2014-08-25 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCP and Patient inclusion: HCP inclusion - HCP Experience with treatment of patients with study compound who have been exposed to risk minimization tools
  Patient inclusion - Patients treated with study compound as per label who have been exposed to the risk minimization materials
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab

SUMMARY:
To evaluate the effectiveness of the YERVOY® educational Risk Minimization (RM) tools in terms of awareness about these tools, their utilization, knowledge and comprehension of Immune Related Adverse Reaction (irAR)s, and appropriate behavior by Healthcare Professional (HCP)s and patients

DETAILED DESCRIPTION:
A total sample size of 160 to 200 HCPs and 160 to 200 patients

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* HCP experienced in the treatment of patients with the research compound and patients that have received at least one dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCPs and Patients in EU member states where YERVOY has been marked for atleast six months
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The proportion of YERVOY HCPs that are aware of the existence of the risk communications tools and how the tools were accessed (i.e. paper or electronic versions) | 6 months
  Distribution metrics and awareness of the tools from responses through the survey will be analysed and descriptive statistics will be used within the different participant groups
Questionnaire: "Who uses the RM communication tools, how, when they are used and how often they are used" | 6 months
  Web downloads metrics will be collected and the usage of tools from responses in the survey will be analysed, and descriptive statistics will be used within the participant groups
Level of knowledge and comprehension of the key elements of important identified risks associated with YERVOY treatment based on the scores obtained from the Questionnaire Surveys | 6 months
  Knowledge and comprehension in HCPs and patients, the knowledge surveys will provide the following data
  1. Total number of responses to the question including the proportions of correct answers to questions where appropriate
  2. Number or frequency and proportion of response options selected
  3. Percentage of responses/total responses per option
  4. Mean value and standard deviation (for appropriate questions)
  From the obtained data, Acceptable levels of correct responses will be determined, post data analysis, reporting and discussion with EMA, to set baseline levels for potential future evaluations and then the scores will be assessed
HCP and patient behaviours via behavioural questions and scenarios based on the scores obtained from the Questionnaire Surveys | 6 months
  For determining appropriate behaviours in HCPs and patients, ideal expected behaviours will be mapped to the ideal care pathway from the Failure Modes and Effects Analysis (FMEA) as described in the RMP. The metrics will show:
  1. Total of number of participants answering the question.
  2. Proportions of participants providing correct answers (to identify knowledge and comprehension)
  3. Proportion of participants showing expected (ideal) behaviour - i.e. correct answers to individual questions.
  4. Proportion of participants showing non-ideal behaviour - i.e. partially correct or incorrect answers to individual questions.
  Analysis will examine knowledge, comprehension and behaviours for different participant types (HCP, Hospital type and Country)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Bristol-Myers Squibb, Princeton, New Jersey, United States
- Local Institution, St Ives, Cambridgeshire, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx